CLINICAL TRIAL: NCT03476681
Title: Phase 1/2 With Expansion Cohorts in a Study of NEO-201 in Adults With Chemo-Resistant Solid Tumors
Brief Title: Study of NEO-201 in Solid Tumors Expansion Cohorts
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Precision Biologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-1801
Record Dates: First submitted 2018-02-26; First posted 2018-03-26 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Cervical Cancer; Uterine Cancer
Keywords: NEO-201; Monoclonal Antibody; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Cervical Cancer; Uterine Cancer; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms; Uterine Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: In the dose expansion phase subjects with non small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), cervical and uterine cancers will be treated with NEO-201 at 1.5 mg/kg every 2 weeks in combination with pembrolizumab at 400 mg IV every 6 weeks.
  In each cycle the combination will be given sequentially with NEO-201 on Day 1, followed by pembrolizumab on Day 2 to reduce the risk of additive infusion reactions. NEO-201 will be administered IV every 2 weeks on Days 1, 15 and 29 of a 42-day cycle.
  Response assessment will be done at the end of Cycle 2 Day 84.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NEO-201 in combination with pembrolizumab (Experimental): Subjects will receive 3 doses NEO-201 in combination with one dose of pembrolizumab in a 42 day cycle. This course will be repeated in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: NEO-201 in combination with pembrolizumab

INTERVENTIONS:
Drug: NEO-201 in combination with pembrolizumab — NEO-201 will be given intravenously every 2 weeks in combination with pembrolizumab. In each cycle subjects will receive 3 doses of NEO 201 and one dose of pembrolizumab.
  Other Names: IHC screening for NEO-201 target

SUMMARY:
The open label, first-in-human, phase 1, dose escalation component in refractory solid tumors has been completed. The Maximum Tolerated Dose and Recommended Phase 2 Dose (RP2D) was determined to be 1.5mg/kg.

The Expansion Phase of this study is currently enrolling subjects with non small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), cervical and uterine cancers who progressed on front line therapy. Subjects will be treated with NEO-201 at the RP2D (1.5 mg/kg) every 2 weeks in combination with pembrolizumab, given 1 day after the NEO-201, at 400 mg IV every 6 weeks.

DETAILED DESCRIPTION:
The experimental drug called NEO-201 (the "study drug") is a monoclonal antibody that is being tested and is not approved for use in the United States by the FDA.

As stated above the RP2D was determined at 1.5 mg/kg and in the current Expansion Phase it will be administered in combination with pembrolizumab. .

A safety lead in will be conducted in the first 3 to 6 subjects to evaluate toxicity prior to expanding accrual. The safety lead-in will be 42 days in length, consisting of 1 dose of pembrolizumab and 3 doses of NEO-201 followed by a 2-week assessment for safety, in subjects with any of the expansion cohorts' targeted disease types. The third patient in the safety lead in must complete the 30-day assessment (1 dose of pembrolizumab and 3 doses of NEO-201 followed by a 2-week safety evaluation) and be evaluated for toxicity prior to treating additional patients.

Following completion of the lead-in, expansion cohorts will accrue subjects with NSCLC, HNSCC, cervical and uterine cancers who progress on frontline therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: >/=18 years
* Diagnosis:

  * Subjects must have histologically or cytologically confirmed recurrent, locally advanced unresectable or metastatic cancer confirmed by the Laboratory of Pathology, NCI
  * Subjects enrolled in the expansion cohorts must have advanced non-small cell lung cancer, HNSCC, uterine cancer, or cervical cancer that has progressed during or after at least one front-line standard of care treatment, including chemotherapy and/or targeted therapy
  * Tumor is positive for NEO-201 antigen expression (defined as at least 10% of tumor cells expressing NEO-201 target antigen).
  * Patient is not a candidate for potentially curative surgery or radiation.

Tumor has the additional characteristics described below for the disease specific expansion cohorts:

NSCLC:

* Tumor(s) must express PD-L1 (TSP > 1%) as determined by an FDA-approved test and/or is microsatellite instability-high (MSI-H) or mismatch repair deficient, and/or is tumor mutational burden-high (TMB-H) [≥10 mutations/megabase (mut/Mb)], as determined by an FDA-approved test.
* Patients with EGFR, ALK1, ROS1 or BRAF V600E genomic tumor aberrations must have had disease progression on FDA-approved agents for these aberrations.
* Patients without these genomic tumor aberrations must have received immune-checkpoint inhibitor previously, either as a single agent or in combination with chemotherapy.

Cervical Cancer:

• Tumor(s) express a combined positive score (CPS) > 1, as determined by an FDA approved test and/or is microsatellite instability-high (MSI-H) or mismatch repair deficient, and/or is tumor mutational burden-high (TMB-H) [≥10 mutations/megabase (mut/Mb)], as determined by an FDA-approved test

HNSCC • Patients are allowed to have received pembrolizumab previously, either alone or as part of a multiagent regimen.

Uterine carcinoma

• Patients who are eligible to have received the combination of pembrolizumab plus lenvatinib (i.e. patients with tumors that are not MSI or dMMR) must have received this regimen, unless considered unsafe due to comorbid conditions (e.g. hypertension, proteinuria).

* Must have archived tissue (10 unstained slides or tissue block), or must have tumor which can be safely biopsied percutaneously and be willing to undergo a tumor biopsy
* MEASURABLE/EVALUABLE DISEASE: Measurable disease (by RECISTv1.1)
* INFORMED CONSENT: Voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care
* PERFORMANCE STATUS: ECOG ≤ 2; or Karnofsky performance status of ≥ 50%
* LABORATORY FUNCTION:

  * Screening laboratory data within 21 days of the first dose of study drug. Subject must have adequate organ function:
  * Hemoglobin > 9 g/dL, or on stable doses (hematocrit stable within 1 gram and dose stable for one month) of erythropoietin or similar medication
  * Absolute neutrophil count (ANC) ≥1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Total bilirubin ≤ 2.0 mg/dL
  * ALT and AST ≤ 3 times the ULN, or, if the subject has liver metastases, ≤ 5 times the ULN
  * Creatinine ≤ 1.5 mg/dL or creatinine clearance > 40 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula
* PRIOR THERAPY:

  * At least 14 days must have elapsed since treatment with oral tyrosine kinase inhibitors, or until toxicities associated with TKI therapy have resolved
  * At least 21 days must have elapsed since treatment with previous monoclonal antibodies, or until toxicities associated with mAb therapy have resolved
  * At least 4 weeks must have elapsed since any chemotherapeutic agents at the time of enrollment (or 6 weeks for regimens containing BCNU or mitomycin C)
  * At least 2 weeks must have elapsed since any systemic corticosteroids at the time of enrollment
  * Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
  * XRT: At least 7 days after local palliative XRT (small port)
* Subjects must have recovered from any acute toxicity related to prior therapy, except for alopecia. Toxicity should be ≤ grade 1, or ≤ grade 2 for peripheral neuropathy, or hypothyroidism
* Subject is expected to be able to remain on a study protocol for at least 8 weeks
* BIRTH CONTROL: Female subject is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study, and 2 weeks after completion of NEO-201 administration or 4 months after the last dose of pembrolizumab (according to package labeling), whichever is later.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 2 weeks after completion of NEO-201 administration or 4 months after the last dose of pembrolizumab (according to package labeling), whichever is later.

Exclusion Criteria:

* History of disseminated or uncontrolled brain metastases or central nervous system disease. Brain metastases will be considered controlled if SD on two consecutive brain MRIs, performed at least 2 months apart, and subject is without seizures.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to NEO-201 or other agents used in this study.
* Any major surgery within 14 days of enrollment.
* Receiving any other investigational agents.
* No archival tissue available and a lesion(s) that cannot be safely biopsied via percutaneous route, or is unwilling to undergo biopsy.
* Has an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, uncontrolled diabetes mellitus, symptomatic congestive heart failure, unstable angina pectoris, hypokalemia, family history of Long QT Syndrome or presence of cardiac arrhythmia.
* Subjects who are assessed to have unacceptable risk of developing infection from neutropenia will be excluded at the Investigator's discretion.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the unknown potential for pharmacokinetic interactions with NEO-201. In addition, these subjects are at increased risk of lethal infections which could complicate the toxicity assessment of this study. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Subject has other serious medical illness, including a second malignancy, or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects due to NEO-201 is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with NEO-201, breastfeeding should be discontinued if the mother is treated with NEO-201.

Additional Exclusion Criteria for Expansion Cohorts

Because patients in the expansion cohort will be receiving pembrolizumab, the following additional exclusion criteria apply:

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to start of study therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Subjects who experienced severe or life-threatening immune-related AEs with prior immune checkpoint therapy requiring medical intervention (steroid or immunosuppressant drugs) and permanent discontinuation of therapy, will be excluded. These include, but not limited to colitis, autoimmune hepatitis, hypophysitis, hyperthyroidism, nephritis, myocarditis, GBS, encephalitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of the combination of NEO-201 with pembrolizumab the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | 1.5 years
  To evaluate toxicity a safety lead in of 3 to 6 subjects will be conducted. The safety lead in will be 42 days long, consisting of 3 doses of NEO-201 and 1 dose of pembrolizumab followed by a 2 week assessment.
  All appropriate treatment areas will have access to a the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm.
Determine Objective Response Rate (either Complete Response or Partial Response) as determined by RECIST v1.1 guidelines | 1.5 years
  For the purposes of this study, subjects will be re-evaluated for response every 12 weeks.
  Response will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Determine Progression Free Survival as determined by RECIST v1.1 guidelines | 1.5 years
  For the purposes of this study, subjects will be re-evaluated for progression every 12 weeks.
  Progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.

SECONDARY OUTCOMES:
Toxicities including treatment emergent adverse events and the character and incidence of Grade 1-4 toxicities. | 1.5 years
  • Describe the character and incidence of Grade 1-4 toxicities based on CTCAE v5.0 that occur in adults receiving NEO-201 in combination with pembrolizumab.
Characterize the area under the concentration-time curve (AUC) of the pharmacokinetics (PK) of NEO-201 combination therapy with pembrolizumab. | 1.5 years
  Quantifiable samples will be drawn at the following time points (during the first 2 Cycles, each Cycle is 42 Days) from the first 6 patients who consent.
  * Cycle1 Day1 (pre dose)
  * 1 hour post dose 1, Cycle1 Day1
  * 4 hours post dose 1, Cycle1 Day1
  * Cycle1 Day2
  * Cycle1 Day4
  * Cycle1 Day6
  * Cycle1 Day8
  * Cycle1 Day15 (pre dose)
  * Cycle2 Day1 (pre dose)
  * 1 hour post dose, Cycle2 Day1
  * 4 hours post dose, Cycle2 Day1
  * Cycle2 Day2
  * Cycle2 Day4
  * Cycle2 Day6
  * Cycle2 Day8
  * Cycle2 Day15 (pre dose)
Characterize Peak Plasma Concentration (Cmax) of the pharmacokinetics (PK) of NEO-201 in combination with pembrolizumab. | 1.5 years
  The reported maximum plasma concentration (Cmax) (Peak concentration) will be determined using a precise validated Elisa method for each dose level on samples collected at the following time points (during the first 2 Cycles, each Cycle is 42 Days)
  * Cycle1 Day1 (pre dose)
  * 1 hour post dose 1, Cycle1 Day1
  * 4 hours post dose 1, Cycle1 Day1
  * Cycle1 Day2
  * Cycle1 Day4
  * Cycle1 Day6
  * Cycle1 Day8
  * Cycle1 Day15 (pre dose)
  * Cycle2 Day1 (pre dose)
  * 1 hour post dose, Cycle2 Day1
  * 4 hours post dose, Cycle2 Day1
  * Cycle2 Day2
  * Cycle2 Day4
  * Cycle2 Day6
  * Cycle2 Day8
  * Cycle2 Day15 (pre dose)
Characterize the Minimum Plasma Concentration (Cmin) of the pharmacokinetics (PK) of NEO-201 in combination with pembrolizumab. | 1.5 years
  The reported minimum plasma concentration (Cmin) (Trough concentration) will be determined using a precise validated Elisa method for each dose level on samples collected at the following time points (during the first 2 Cycles, each Cycle is 42 Days).
  * Cycle1 Day1 (pre dose)
  * 1 hour post dose 1, Cycle1 Day1
  * 4 hours post dose 1, Cycle1 Day1
  * Cycle1 Day2
  * Cycle1 Day4
  * Cycle1 Day6
  * Cycle1 Day8
  * Cycle1 Day15 (pre dose)
  * Cycle2 Day1 (pre dose)
  * 1 hour post dose, Cycle2 Day1
  * 4 hours post dose, Cycle2 Day1
  * Cycle2 Day2
  * Cycle2 Day4
  * Cycle2 Day6
  * Cycle2 Day8
  * Cycle2 Day15 (pre dose)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Conlon, MD, Principal Investigator — National Cancer Institute - Women's Malignancy Branch; Azam Ghafoor, MD, Principal Investigator — National Cancer Institute - Thoracic and GI Malignancy Branch; Charalampos Floudas, MD, Principal Investigator — National Cancer Institute - Head and Neck/GUMB
Locations (2):
- United States (2):
  - National Cancer Institute, Bethesda, Maryland
  - INOVA Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cole CB, Morelli MP, Fantini M, Miettinen M, Fetsch P, Peer C, Figg WD, Yin T, Houston N, McCoy A, Lipkowitz S, Zimmer A, Lee JM, Pavelova M, Villanueva EN, Trewhitt K, Solarz BB, Fergusson M, Mavroukakis SA, Zaki A, Tsang KY, Arlen PM, Annunziata CM. First-in-human phase 1 clinical trial of anti-core 1 O-glycans targeting monoclonal antibody NEO-201 in treatment-refractory solid tumors. J Exp Clin Cancer Res. 2023 Mar 29;42(1):76. doi: 10.1186/s13046-023-02649-6. PMID 36991390